CLINICAL TRIAL: NCT05301829
Title: Thrombin Generation Assay to Assess Thrombotic Risk and the Evolution of the Hypercoagulability Profile of Patients With Nephrotic Syndrome
Brief Title: Thrombin Generation Assay to Assess Thrombotic Risk in Nephrotic Patients
Acronym: TGANephrotic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220213
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic Syndrome; Thrombotic risk assessment
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of citrated whole-blood samples three times during the timecourse of the disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The thromboembolic risk is increased during the nephrotic syndrome (NS) with an incidence of deep vein thrombosis 15%, pulmonary embolism of 10-30% and renal vein thrombosis of 25-37%. There is a hemostatic imbalance with urinary leakage of anticoagulant factors and increased hepatic synthesis of procoagulant factors, platelet hyperaggregability and a decrease in fibrinolytic activity. However, the identification of patients requiring anticoagulant prophylaxis remains imprecise.The thromboembolic risk is higher when the NS is related to extramembranous glomerulonephritis comparatively to others glomerulopathies. The reason of this difference is not still known. This risk increase with SN's severity and therefore with the decrease of albuminemia. Moreover, few studies have evaluated anticoagulant treatment efficacy during a NS, which clinical benefit depends also on hemorrhagic risk specific of each patient. Thus, the determination of the thrombotic risk and the modalities of anticoagulation are variable and perfectible during the NS.

We propose to use the thrombin generation test (TGT) to quantify the thromboembolic risk in patients with a NS and to follow its evolution during prophylactic anticoagulation and after remission of NS.

DETAILED DESCRIPTION:
Thrombin generation test will be performed prospectively in nephrotic patients with various diseases (Minimal Change Disease (MCD), Malignant Nephrosclerosis (MN), Focal Segmental GlomeruloSclerosis (FSGS), diabetic glomerulopathy…) at diagnosis, during anticoagulant treatment (D8±3) and after disease remission (M6).

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic syndrome
* Known cause of nephrotic syndrome (renal biopsy and/or positive anti-PLA2R)

Exclusion Criteria:

- Active anticoagulation treatment before TGT

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with nephrotic syndrome defined by albuminemia <3 g/dl and urinary protein/creatinine > 3g/g) admitted in the nephrology department of Tenon hospital; etiological diagnosis available; consenting to research and whose treatment and follow-up will be possible for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the prognosticity of TGT in predicting the occurrence of a thromboembolic event at 6 months. | 6 months
  Number of thrombotic events at 6 months of follow-up

SECONDARY OUTCOMES:
Variation of TGT parameters (data combined considering latency, velocity, peak, amount of total thrombin formed) during the follow-up | Maximum 6 months (when albumin > 30 g/l)
  To calculate the difference of TGT parameters between the time of acute phase of NS (at diagnosis = inclusion), and after NS remission.
Compare the theoric indications for anticoagulation therapy according to TGT parameters with those of the Lin R algorithm and "Kidney Disease: Improving Global Outcomes" (KDIGO) 2021 | At diagnosis = at inclusion
  Percentage of anticoagulated patients versus theoric number, based on TGT results and available algorithms

CONTACTS AND LOCATIONS:
Overall Officials: Armance MARCHAL, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Néphrologie et Dialyses, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided